CLINICAL TRIAL: NCT00517972
Title: Omacor for Perimenopausal Depression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Reliant Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC#06-102;IND76801
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: perimenopausal depression; omacor; major depressive disorder; women
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Omacor (omega-3-acid ethyl esters)

SUMMARY:
Recently, antidepressants and other similar acting agents have been explored as a class of medications to treat major depressive disorder (MDD) in the context of perimenopause, as well as the somatic symptoms of perimenopause (such as hot flashes). Omega-3 fatty acids, which include eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), are nutritional compounds with widely established health benefits and which occur naturally in fish and marine sources. Results of previous mood disorder studies have indicated that omega-3 fatty acids may be of help in the treatment of depression. Therefore, the current study is designed to examine the effectiveness and tolerability of the study drug, Omacor, (omega-3 fatty acid ethyl esters), in the treatment of major depressive disorder in perimenopausal women.

DETAILED DESCRIPTION:
Over twenty percent of women will experience a major depressive episode in their lifetimes, a prevalence that reflects a greater risk than is found among men. Perimenopause is commonly defined as a time of hormonal fluctuation that typically occurs in women 40-55 years of age with changes in menstrual patterns. It has been demonstrated that women may be at a particularly high risk for depressive symptoms during perimenopause. Hormone replacement therapy, particularly estrogen, may help with mood symptoms in the perimenopause. However, hormone replacement therapy (HRT) has become increasingly controversial in light of the findings of the Women's Health Initiative study. In that study, HRT was associated with an increased risk of some serious health problems without many of the benefits which had been previously attributed to HRT. Since the report of these results, HRT use has declined and other agents such as antidepressants have been used as an alternative treatment for depression in perimenopausal women.

Optimal treatments for depression must be safe and effective, with ideal treatments also providing other health benefits as well. Omega-3 fatty acids are nutritional compounds with widely established health benefits. Eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are omega-3 fatty acids found in fish and marine sources. Mood disorder studies have supported a role for omega-3 fatty acids in the treatment of depression. In a study from 1998, it was demonstrated in a cross-national study that the risk of major depression is inversely associated with per capita fish consumption. Several other studies have demonstrated that in depressed subjects, there is a lower total omega-3 fatty acid content in the membranes of red blood cells and plasma (liquid part of the blood) when compared to control subjects. Treatment data from studies of major depressive disorder also support a role for omega-3 fatty acids, especially when omega-3 fatty acids are used as an adjunctive treatment, i.e., fatty acids are administered along with another therapeutic compound during treatment of major depressive disorder.

It has also been demonstrated that the use of antidepressants such as fluoxetine, paroxetine, and venlafaxine for treatment of hot flashes and citalopram for the treatment of hot flashes and mood in perimenopausal women are more effective than placebo. However, antidepressant medications are associated with significant side effects and as of late, have come under increased scrutiny by the U.S. FDA, the psychiatric, and general medical community due to the ongoing controversy regarding a possible increased risk of suicidality after the initiation of antidepressant treatment. While there is not complete agreement on the mechanism of action for omega-3 fatty acids, like antidepressants, overall data suggests that omega-3 fatty acids may be beneficial for treatment of perimenopausal depression. However, unlike antidepressants, omega-3 fatty acids are naturally occurring substances, which may appeal to many individuals suffering from perimenopausal depression. Omega-3 fatty acids have known benefits for cardiovascular health. Therefore, the current study is designed to examine the effectiveness and tolerability of the study drug, Omacor, (omega-3 fatty acid ethyl esters), in the treatment of major depression in perimenopausal women.

Subjects that take part in this voluntary study will undergo 6 clinic visits during the 8-week study period. The first visit may last up to 3 hours, with all other clinic visits lasting approximately 45 minutes. Once the consent form has been read and signed, subjects will be enrolled in the study. At the first visit, medical and psychiatric histories will be reviewed. All participants will undergo the standardized protocol for establishing depression, the Structured Clinical Interview for DSM-IV (SCID), in addition to being rated by symptom rating scales that include the Clinical Global Impression (CGI) and the Hamilton Depression Rating Scale (HAM-D (17-item). All participants will also undergo an entry interview that will include a psychiatric and substance use history (including data regarding use of alcohol, tobacco, and illicit substances). During the initial exam, vital signs (height, weight and blood pressure) will also be recorded for all participants. In addition, all subjects that are enrolled must have had a gynecologic exam within the past year, or if not, will be given a referral for such an exam. Blood (approximately 3 teaspoons) will be drawn for routine laboratory testing (thyroid function tests (TFTs) and complete blood count (CBC)) and a lipid profile. Blood will also be drawn (approximately 3 teaspoons) at the last visit for the purpose of repeating the lipid profile. Subjects will also complete the Greene Climacteric Scale (GCS), which is used to quantify the severity of perimenopausal somatic symptoms, including hot flashes.

As this study will be examining omega-3 fatty acids, subjects will not be eligible to participate in the study if they are taking omega-3 fatty acid supplements. In addition, once enrolled in the study, all participants will be asked to avoid taking additional omega-3 fatty acids or enhanced food products and will need to avoid increasing or decreasing the amount of fish that they normally eat during the entire time of the study.

Once all interviews and medical screens are finished, all participants will receive the study medication (Omacor). The study drug will be supplied in 1 gram capsules and participants will need to take two capsules at the same time every day. Thus, all subjects will be taking a total of 2 grams of Omacor per day.

Questions about mood and perimenopausal symptoms will be asked at each visit. At each of these visits, the primary efficacy measures (CGI, HAM-D, and GCS) will be administered. The GCS will be completed at each visit to quantify the somatic symptoms of perimenopause. Subjects will also be asked the about number of missed doses each week.

Telephone contact with investigators is permissible and will be available 24 hours/day for emergencies. All contacts will be documented in the participant's records.

ELIGIBILITY:
Inclusion Criteria:

* Women age 40 years old or older.
* Subjects must have perimenopausal symptoms of at least 3 months duration, and which include irregular periods and/or hot flashes.
* Subjects must have a minimum score of 15 on the Hamilton Rating Scale for Depression.
* Subjects must be willing to be treated on an outpatient basis.
* Subjects must provide written informed consent.

Exclusion Criteria:

* Subjects presently taking antidepressant medication.
* Subjects currently using hormone replacement therapy (HRT).
* Subjects currently taking omega-3 fatty acid supplements.
* Presence of psychotic symptoms.
* History of mania or hypomania.
* Hamilton Rating Scale for Depression (HAM-D) suicide item score > 3.
* Abnormal uterine bleeding (heavy or prolonged uterine bleeding, menstrual periods occurring more frequently than every 3 weeks, bleeding after sexual intercourse, spotting between periods) that has not been evaluated by a gynecologist.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Reduction of the initial HAM-D score by 50% or more at week 8 of the trial.
Reduction of the HAM-D score to less than 7 at week 8.
Clinical Global Impression change in score achievement to "very much improved" or "much improved" at week 8.

SECONDARY OUTCOMES:
Decrease in the Greene Climacteric Scale by 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P Freeman, M.D., Principal Investigator — University of Arizona
Locations (1):
- Women's Mental Health Program; University of Arizona, Tucson, Arizona, United States